CLINICAL TRIAL: NCT00630890
Title: Phase I Dose Escalation Trial of External Beam Radiation and Cyberknife Radiosurgery Boost With Concurrent Capecitabine for Hilar Cholangiocarcinoma (Klatskin Tumor)
Brief Title: Cyberknife Radiosurgery Boost for Hilar Cholangiocarcinoma (Klatskin Tumor)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: investigator left UCSF and study was closed prematurely in 2008. No results to report.
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07455
Record Dates: First submitted 2008-02-28; First posted 2008-03-07 (Estimated); Last update posted 2015-09-11 (Estimated); Status verified 2015-09

CONDITIONS: Cholangiocarcinoma; Klatskin Tumor; Biliary Tract Cancer
Keywords: Hilar Cholangiocarcinoma (Klatskin Tumor); External Beam Radiation; Cyberknife; Capecitabine
MeSH Terms: conditions — Cholangiocarcinoma; Klatskin Tumor; Biliary Tract Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): External beam radiation with Cyberknife radiosurgery boost and concurrent capecitabine
  Interventions: Radiation: External beam radiation and Cyberknife radiosurgery boost and capecitabine

INTERVENTIONS:
Radiation: External beam radiation and Cyberknife radiosurgery boost and capecitabine — External Beam Radiation to 45 Gy Stereotactic Body Radiotherapy with Cyberknife to 20 Gy in 5 fractions dose escalation to 25 Gy in 5 fractions, and then 30 Gy in 5 fractions Capecitabine 825 mg/m2 q12 hours taken orally 5 days per week
  Other Names: Xeloda

SUMMARY:
The purpose of this study is to test the safety of giving external beam radiation, followed by a Cyberknife radiosurgery boost at different dose levels, together with a chemotherapy drug called capecitabine. The dose of Cyberknife radiosurgery boost will be made higher slowly in this protocol. Patients with hilar cholangiocarcinoma (Klatskin tumor), which is not amenable for surgical removal, are eligible.

The hypothesis is that highly focused high dose radiation delivered using Cyberknife in conjunction with traditional radiation and chemotherapy can improve outcome in this patient population.

DETAILED DESCRIPTION:
This is a dose escalation study which will escalate the dose of Cyberknife radiosurgery boost after external beam radiation of 45 Gy with concurrent capecitabine. The three dose levels are 4 Gy x5, 5 Gy x5 and 6 Gy x 5, with 3 patients at each dose level. Dose-limiting toxicity (DLT) is defined as acute grade 3 liver or intestinal toxicity or any acute grade 4 toxicity. If one patient experienced a DLT at a particular dose level, the cohort should be expanded to 6 patients. The maximum tolerated dose (MTD) is defined as the dose level below that which results in DLT in 2 or more of the 6 patients in each cohort. At least 5 patients should be enrolled in the cohort of 6 Gy x 5 even if none of the first 3 experienced DLT, as a means of added verification of dose tolerance, at this upper limit of dose for this study.

The patient population includes any patients who have unresectable hilar cholangiocarcinoma without any prior history of radiation. We anticipate accruing 1 patient every 2 months; therefore, we estimate that it will require approximately 22 months to accrue 11 patients if no DLT is experienced by any patients requiring expansion of the cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Age eighteen years or older
* Histological defined unresectable cholangiocarcinoma of hilar region of the liver
* Patients should have evaluable disease on one or more imaging modalities (CT scan, MRI, and/or PET) since this will be necessary for radiation treatment planning. However, because the borders of these tumors are sometimes difficult to define precisely, measurable disease is not required (see Section 9.1 for definitions of evaluable and measurable disease).
* The maximum tumor dimension should be less than 6 cm.
* Patients with pathologically enlarged perihepatic regional lymph nodes are allowed.
* Prior surgical resection is allowed if there is gross disease remaining
* Adjuvant chemotherapy is allowed at least 1 month after completion of radiation therapy if any grade 3 or higher toxicity has resolved
* Percutaneous biliary drains and biliary stents are allowed
* Performance status of ECOG 0-1 (see Appendix I)
* Life expectancy greater than 6 months
* Subject must have normal organ and marrow functions as defined below

  * leukocytes >3,000/mcL
  * absolute neutrophil count >1,500/mcL
  * platelets >100,000/mcL
  * total bilirubin <2.5 X institutional upper limit of normal
  * AST(SGOT)/ALT(SGPT) <2.5 X institutional upper limit of normal
  * creatinine within normal institutional limits OR
  * creatinine clearance >60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal.
  * PT/PTT within normal institutional limits
* Gold marker seeds (1 to 3) are required to be placed in or around the primary tumor by an interventional radiologist
* Ability to give written informed consent and willingness to comply with the requirements of the protocol
* Women of child-bearing potential must agree to use an effective method of birth control during treatment and for six months after receiving their last dose of treatment

Exclusion Criteria:

* Patients who have had prior chemotherapy
* Patients who have had external beam radiation to the region of liver hilar previously.
* Patients receiving any other investigational agents
* Patients with known metastases
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to capecitabine.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients who are not candidates for gold marker seeds placement due to position of the tumor or co-existing medical condition.
* Pregnant or lactating women and women of child-bearing potential who are not using an effective method of birth control
* Any condition that compromises compliance with the objectives and procedures of this protocol, as judged by the principal investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2007-10; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
To evaluate acute toxicities | 3 months for acute toxicities
To determine the maximal tolerated dose of the Cyberknife radiosurgery boost | 3 months for acute toxicities

SECONDARY OUTCOMES:
To assess local and regional control | two years
To evaluate radiographic response | two years
To assess delayed and long-term toxicities | two years
To estimate disease specific and overall survival | two years

CONTACTS AND LOCATIONS:
Overall Officials: Kim Huang, M.D., Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States